CLINICAL TRIAL: NCT03388372
Title: Efficacy and Safety of Nimotuzumab in Addition to Radiotherapy and Temozolomide for Cerebral Glioblastoma
Brief Title: Nimotuzumab Plus Radiotherapy With Concomitant and Adjuvant Temozolomide for Cerebral Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shao Xiong Wu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NimotuzumabGBM2010
Record Dates: First submitted 2017-12-11; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Glioblastoma
Keywords: glioma; phase 2; nimotozumab; temozolomide; radiotherapy
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — nimotuzumab; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab plus RT and temozolomide. (Experimental): Nimotuzumab, administered once a week intravenously in addition to radiotherapy with concomitant and adjuvant temozolomide (TMZ) after surgery.
  Interventions: Biological: Nimotuzumab; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Biological: Nimotuzumab — Nimotuzumab, 200 mg as 1-hour intravenous infusion once weekly, from first week to last week of RT for a total of 6 times.
Drug: Temozolomide — Temozolomide, 75 mg/m2/d was administered orally from the first to the last day of RT. After 4-week break, individualized adjuvant TMZ was given based on MGMT status. The standard 5-day schedule every 4 weeks for six cycles was given for patients with negative MGMT expression. Dose was 150mg/m2 for the first cycle and 200 mg/m2 from the second cycle. The 7-day on/7-day off schedule every 2 weeks for 12 cycles was given for patients with positive MGMT expression. The dose was 100 mg/m2 for the first two cycles and 150 mg/m2 starting from the third cycle.
Radiation: Radiotherapy — Fractionated 3D conformal RT was given at 2.0Gy per fraction, 5 daily fractions per week for 6 weeks.

SUMMARY:
This study aimed to investigate the clinical benefit contribution and safety of nimotuzumab to the standard combined treatment for patients with newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically proven single supratentorial GBM (WHO grade 4);
* EGFR positive;
* >50％ of the gross tumor volume removed by surgery；
* Karnofsky performance score (KPS) ≥ 60;
* Adequate renal function (creatinine ≤1.5×upper limit of normal [ULN] or creatinine clearance ≥ 60 mL/min), hepatic function (total bilirubin ≤1.5×ULN and serum transaminases ≤3×ULN), and hematologic function (white blood cell count ≥ 3,000/uL or absolute neutrophil count ≥ 1,500/uL, platelets ≥ 100,000/uL, and hemoglobin ≥ 10 g/dL).
* Tumor tissue was required for central pathology review and re-checking EGFR and MGMT expression status;
* An interval of 2 to 6 weeks between surgery and RT was required.

Exclusion Criteria:

* Negative EGFR expression;
* Prior chemotherapy, anti-EGFR therapy, RT, or a history of malignancy in the previous 5 years;
* Patients with severe complications or active infection;
* Continuous vomiting that could interfere with the oral administration of TMZ;
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-08-18 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS will be calculated as the time from surgery to the date of progression-free.
Overall survival (OS) | 2 years
  OS will be calculated as the time from surgery to the date of death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR: overall response rate (ORR), subjects will be classified according to the RANO criteria, which is a composite of MRI changes, clinical response and changes in steroid use.
Incidence of adverse events | 6 months
  Incidence of adverse events.Toxicities will be tabulated and graded according to the NCI Common Toxicity Criteria (CTCAE) version 3.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Xiong Wu, Professor, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Brain Hospital, Guangdong
  - The First Affiliated Hospital/School of Clinical Medicine of Guangdong, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Shenzhen People's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided